CLINICAL TRIAL: NCT06271044
Title: Reducing Radioiodine Treatment in Low Risk Papillary Thyroid Cancer
Brief Title: a. Reducing Radioiodine Treatment in Papillary Thyroid Cancer. RAILESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paivi Halonen, Medical Oncologist, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RAILESS
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: to Omit Radioiodine Treatment Safely in Patients With Low -Risk Papillary Thyroid Cancer With Seize of 11-20mm
Keywords: radioiodine treatment, low risk thyroid cancer, papillary thyroid cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Intervention Model Description: Patients with low risk papillary thyroid cancer either received a radioiodine treatment according to the normal Finnish treatment schedule or were schedulded for only follow-up .
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAILESS (No Intervention): Railess group including patients to bw followed up wihtout postoperative radioiodine treatment
- rairinn (Active Comparator): THose patients receiving radioiodine treatment according to the normal treatment practice at that time
  Interventions: Other: With radioiodine treatment; Procedure: With postoperative radioiodine treatment

INTERVENTIONS:
Other: With radioiodine treatment — Postoperative radioiodine not given
  Other Names: RAILESS
  Arms: rairinn
Procedure: With postoperative radioiodine treatment — Postoperative radioiodine given
  Other Names: RAIRINN
  Arms: rairinn

SUMMARY:
To study if its is safe to reduce the amount of postoperative treatments in those patients, who have been operated on because of a low-risk intrathyroidal papillary thyroid cancer with diameter of 11-20mm, and in whom postoperative thyroglobulin levels are of low level.

DETAILED DESCRIPTION:
The purpose of the study : to enroll about 50 patients operated on because of a low-risk intrathyroidal papillary thyroid cancer with diameter of 11-20mm, and in whom postoperative thyroglobulin levels are of low level.

Methods: either to follow-up patients according to the study protocol without radioiodine treatment or to give a radioiodine treatment with a dose of 1.1 GBq according to the normal Finnish treatment protocol for papillary thyroid cancer to those patients who themselves preferred to have a normal postoperative treatment.

ELIGIBILITY:
Inclusion Criteria:

* low risk papillary intrathyroidal thyroid cancer with diameter of 11-20mm
* no lymphnode metastases

Exclusion Criteria:

* high risk papillary cancer
* mutlifocal papillary cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event free situation during follow-up event free /disease free | 10 yrs
  Without any treatmment

CONTACTS AND LOCATIONS:
Overall Officials: Päivi Halonen, MD, Principal Investigator — Medical Oncologist

IPD SHARING:
Plan to Share IPD: Undecided